CLINICAL TRIAL: NCT05336136
Title: Custom Non-invasive Ventilation Masks in Children
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alberta (Other)
Collaborators: Stollery Children's Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: Pro00047768
Record Dates: First submitted 2021-06-07; First posted 2022-04-20 (Actual); Last update posted 2025-01-08 (Actual); Status verified 2025-01

CONDITIONS: Noninvasive Ventilation; Child, Only; Adherence, Patient
MeSH Terms: conditions — Patient Compliance

STUDY DESIGN:
Intervention Model Description: Within subject crossover
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Custom mask (Experimental): Custom mask based on 3D facial photograph for administration of non-invasive ventilation
  Interventions: Device: Custom mask
- Current commercial mask (Active Comparator): Current commercial mask used by the participant for administration of non-invasive ventilation
  Interventions: Device: Current commercial mask

INTERVENTIONS:
Device: Custom mask — Custom mask based on 3D facial photograph for administration of non-invasive ventilation
  Arms: Custom mask
Device: Current commercial mask — Current commercial mask used for administration of non-invasive ventilation
  Arms: Current commercial mask

SUMMARY:
One significant challenge to non-invasive ventilation (NIV) use in children is finding masks to fit a wide range of growing shapes and sizes. While the technology has improved with development of masks specifically for children, the range of options remains limited. Given the smaller size relative to adults, craniofacial abnormalities and craniofacial differences are more likely to compromise mask fit for children. A poor mask fit is uncomfortable, alters delivery of airway pressure, and, in some children, leads to failure of NIV and the need for surgical insertion of an airway in the neck to deliver positive airway pressure through a tracheostomy. This makes expanding the technology to deliver NIV vital and custom NIV masks an exciting solution.In this study, this study will enroll children who are established on long-term NIV with at least some use within 3 months of starting this therapy but who have non-optimal adherence. After consenting to participate and completing demographic and health questionnaire, participants will undergo a facial scan using stereophotogrammetry. This scan will be imported into a computer-aided design software to create a NIV mask customized to the individual face. The steps of mask testing will include: i) Bench testing to compare the leak and comfort parameters of the current commercial mask used by the participant to the custom mask: ii) Efficacy of treatment as measured by polysomonography iii) NIV compliance from machine downloads; iv) Questionnaires to assess the subjective comfort, fit, and adverse events Finally, participants and their parents/guardian will be asked which mask they prefer and why.

DETAILED DESCRIPTION:
1. Background 1.1 Investigational Device Custom non-invasive ventilation (NIV) masks will be fabricated based on a facial scan of the participant using sterophotogrammetry (3D photography). The scanner captures and digitizes facial features in a 180o ear-to-ear view in a few seconds. The points in the data set represent the surface of the face. This data set is then converted into a surface representation that can be manipulated using computer-aided design software (MeshMixer, Autodesk, San Rafael, CA). The facial scan data will be imported into computer-aided design (CAD) software (Fusion 360, Autodesk, San Rafael, CA) to create an NIV mask that is customized to the individual face. Once the design is created, a mold will be printed out of polylactic acid filament using a fused filament fabrication 3D printer (Ultimaker II, Ultimaker North America, Cambridge, MA). The printed mold will then be injected with medical grade silicone (Dragonskin, Smooth-On, Macungie, PA), and cured overnight. The coupler, used to attach the mask to the tubing connected to the ventilator, will be directly printed using stereolithography (SL Moai, Peopoly, Los Angeles, CA).

   1.2 Previous Studies and Predicate Devices A few reports indicate that quantitative approaches towards NIV mask selection may improve comfort and adherence to treatment. In 2018 Ma et al. reviewed selection and design considerations for continuous positive airway pressure (CPAP) masks and stated "There is potential for optimizing the CPAP mask fit by adapting the interface to the patients' individual characteristics. This holds particularly true for users with abnormal features or simply outside conventional industry sizing standards. There is to date no integrated system that integrates those elements into a standard solution, but several studies have shown its effectiveness for specific cohorts."1

   In 2019, Goh et al. reported a quantitative analysis of facial photographs of obstructive sleep apnea (OSA) patients.2 This report suggests that quantifying individual craniofacial features may help guide mask choice for NIV treatment for OSA, although the authors cautioned that the oronasal masks were not as effective as the nasal masks in terms of leakage and in reducing the number of apnea events. Despite the caveats, the report supports that further study of aa more rigorous approach to mask fitting is warranted. In an accompanying commentary, Cistulli and Sullivan state: "Surprisingly, the evidence base supporting clinical decisions about appropriate mask selection is relatively weak and is based largely on art rather than science."3

   At least two companies offer custom NIV masks, including Inspirate (Singapore) and ApneaSeal, (Australia). To our knowledge, however, efficacy and compliance of custom versus commercial masks has not been tested rigorously. In addition, the published literature on customized masks for NIV therapy is small. For creating the masks de novo, one report details the fabrication of customized masks using maxillofacial prosthodontic laboratory techniques,4 while another reports a procedure including impression casting, 3D printing and silicone casting.5 Another approach describes modifying standard masks to create 3D-printed interfaces fitted to individual faces.6

   1.3 Trial Conduct This study will be conducted in compliance with the protocol approved by the University of Alberta Health Research Ethics Board (HREB), and according to Good Clinical Practice standards.

   1.4 Population Children already established on NIV (use for at least 3 month) between the ages of 6-12 years who continue to show sub-optimal adherence are able to be the participants in this clinical trial. Children with craniofacial disease or differences make up a large proportion of children using NIV. Craniofacial dimensions change with growth such that children using NIV may need to change to a different mask to provide the best possible fit. Children with developmental or physical disabilities that would prevent their successful completion of the study protocol (e.g., non-verbal, unable to follow 3-step commands, unable to lie still for 20 min) will be excluded from recruitment.
2. Trial Objectives To compare the efficacy of custom NIV masks to commercial masks as measured by efficacy of treatment delivery, compliance, fit test, and ratings of comfort.
3. Trial Design 3.1 Study Design/Type This is a non-randomized clinical trial using a crossover design comparing a custom NIV mask to the participants current commercial NIV mask.

   3.2 Procedures

   There will be three parts to this trial to compare the custom mask to the participant's current commercial mask:

   i) Fit testing will assess both the unintentional leak and comfort of the custom mask compared to the participant's current commercial mask. This will be completed with the participant sitting in a seated position. For each mask, an in-line flow sensor will be used to assess unintentional leak (i.e., air leak around the mask) at two levels of mask tightness (typical used at home, loose) and two pressures (current mean airway pressure, 4 cmH20 higher). Participants will be asked to rate comfort for each trial using a pictorial visual analogue scale. The total testing time including set-up will be approximately 45 min.

   ii) Titration polysomnography will assess the treatment efficacy. Participants will undergo a standard clinical polysomnography in the Pediatric Sleep Laboratory using their current commercial mask and then the custom mask prior with a 2-week measurement of compliance after each polysomnography study. The titration studies will be scored according to the Pediatric Sleep Laboratory protocol and the data extracted for analysis.

   iii) NIV compliance & end of trial questionnaire will assess compliance from NIV machine downloads as well as mask comfort and fit prior to and at the end of each 2-weeks compliance monitoring period, and preference assessed at the end of the study. After each titration study (custom, commercial mask), participants will use the same mask for 2-weeks with NIV machine downloads obtained specific to this time period for each mask. At the end of each 2-week period, participants and their parent/guardian will be asked to complete a questionnaire to assess participantive comfort and fit using a pictorial visual analogue scale as well as to provide narrative data on their experience. Participants and their parent/guardian will also be asked to describe any adverse events. There will be a minimum 2-week wash out period between mask trials where the participants will wear their current commercial ask without monitoring. After each participant has completed both 2-week trials, the participant and their parent/guardian will be asked which mask they prefer and why. The decision as to whether the custom mask is appropriate for on-going use outside the trial will be made by the participant, their parent/guardian, and the NIV clinical team (includes physicians, an NIV nurse practitioner, and an NIV respiratory therapist).
4. Statistical Plan 4.1 Statistical Methods Descriptive statistics will be used to summarize demographic and health information of the participants. Pair-wise t-tests will be used to compare continuous data including unintended air leak, polysomnography variables, and compliance measurements between custom and commercial masks with corrections for multiple comparisons as appropriate. Categorical data, including comfort and mask preference, will be analyzed using Chi-square or Kruskal-Wallis tests.

4.2 Participant Population(s) for Analysis Power calculations show that based on the recruitment of 15 participants, we will have the ability to detect a 1 hour increase in NIV compliance (increase in average use per day from 360 min to 420 min, SD 60 min) with power = 0.86, α = 0.05. Participants will be identified through the NIV clinic and approached for participation as they are identified. As the sample is not random and will focus on those with low compliance, the study results will be relevant to those children most likely to benefit from a custom mask.

ELIGIBILITY:
Inclusion Criteria:

* Children between 8-12 years of age
* Followed clinically by the Non-invasive ventilation clinic at the Stollery Children's Hospital
* Established on non-invasive ventilation as part of their treatment plan.

Exclusion Criteria:

* Children with developmental or physical disabilities that would prevent their successful completion of the study protocol (e.g., non-verbal, unable to follow 3-step commands, unalbe to lie still for 20 min).
* Children whose parent/guardian are unable to provide consent because of an inability to read the study documents in english.

Ages: 8 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 15 (Estimated)
Dates: Start 2023-12-15 (Actual); Primary Completion 2026-01 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Change in apnea hypopnea index | Baseline (commercial mask study), repeated measure at 1 month (custom mask)
  Polysomnography parameter - apnea hypopnea index
Change in obstructive apnea hypopnea index | Baseline (commercial mask study), repeated measure at 1 month (custom mask)
  Polysomnography parameter - obstructive apnea hypopnea index
Change in oxygen desaturation index | Baseline (commercial mask study), repeated measure at 1 month (custom mask)
  Polysomnography parameter - oxygen desaturation index
Change in percent time with oxygen saturation less than 90% | Baseline (commercial mask study), repeated measure at 1 month (custom mask)
  Polysomnography parameter - percent time with oxygen saturation less than 90%
Change in percentage of nights used | Two weeks of commercial versus custom mask use
  Machine download
Change in average time used/night | Two weeks of commercial versus custom mask use
  Machine download

SECONDARY OUTCOMES:
Change in mask air leak (bench testing) | Baseline (commercial mask study), repeated measure at 1 month (custom mask)
  Unintentional mask leak
Change in mask comfort - participant (visual likert scale, 1-9) | End of two week of mask use of commercial versus custom mask
  Subjective rating of mask comfort from participant
Change in mask comfort - parent (visual likert scale1-9) | End of two week of mask use of commercial versus custom mask
  Subjective rating of mask comfort from parent
Mask preference - participant (question) | End of trial - 1 month
  Participant selection of mask preference with reasons
Mask preference - parent (question) | End of trial - 1 month
  Parent selection of mask preference with reasons

CONTACTS AND LOCATIONS:
Overall Officials: Joanna E MacLean, MD, PhD, Principal Investigator — University of Alberta
Locations (1):
- University of Alberta, Edmonton, Alberta, Canada

IPD SHARING:
Plan to Share IPD: No